CLINICAL TRIAL: NCT00795275
Title: Exploring the Incretin Effect in People With IFG
Brief Title: Incretin Effect in People With Impaired Fasting Glucose
Acronym: 1651
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0749
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: pre-diabetes; isotopes; insulin secretion; insulin action; GLP-1; simple obesity; impaired fasting glucose
MeSH Terms: conditions — Obesity; Glucose Intolerance | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Impaired Fasting Glucose (Experimental): Treatment of people with impaired fasting glucose with Januvia (sitagliptin phosphate)
  Interventions: Drug: Sitagliptin Phosphate
- Normal glucose tolerance (Experimental): Treatment of people with normal glucose tolerance with Januvia (sitagliptin phosphate)
  Interventions: Drug: Sitagliptin Phosphate

INTERVENTIONS:
Drug: Sitagliptin Phosphate — Januvia 100 mg po qd x 28 days for all subjects after baseline measures made
  Other Names: brand name: Januvia

SUMMARY:
Regulation of endogenous glucose production (EGP) and insulin secretion are major actions of glucagon-like peptide-1 (GLP-1). Determining whether alterations in GLP-1 may contribute to abnormal EGP and insulin secretion in people with impaired fasting glucose (IFG) was the objective of the current study. The investigators hypothesized that defects in GLP-1 may explain the inappropriate basal EGP and diminished insulin secretion in IFG, and, furthermore, that by increasing circulating GLP-1 levels (using a new medicine called "sitagliptin") the investigators could reverse these defects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, sedentary, non-smokers, men and women 45-70 years old Subjects were placed into 1 of the 2 groups based on two 2-hour 75g oral glucose tolerance tests (2h OGTT), separated by one week: a control group with normal glucose tolerance (NGT; n=14; fasting glucose <5.6 mmol/l and 2h OGTT <7.8 mmol/l), or IFG (n=10; fasting glucose 5.6-6.9 mmol/l, and 2h OGTT <7.8 mmol/l).

Exclusion Criteria:

* Subjects were excluded for: thyroid stimulating hormone <50 or >500 milliunits/L, fasting triglycerides >10.3 mmol/l, creatinine >130 μmol/l, elevated liver function tests (>2 times normal), hematocrit < 38%, or white blood cell count <3.0 x 103. Use of medications for lipid and/or glucose lowering also excluded enrollees. Women may not have used hormone replacement therapy in the past 1 year. Smokers. BMI <25 or >40 kg/m2. Diabetes or impaired glucose tolerance.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Perreault, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perreault L, Man CD, Hunerdosse DM, Cobelli C, Bergman BC. Incretin action maintains insulin secretion, but not hepatic insulin action, in people with impaired fasting glucose. Diabetes Res Clin Pract. 2010 Oct;90(1):87-94. doi: 10.1016/j.diabres.2010.06.012. Epub 2010 Aug 13. PMID 20708814

RESULTS

PARTICIPANT FLOW:
Groups:
- People With Impaired Fasting Glucose: people with impaired fasting glucose
  Januvia (sitagliptin phosphate) : Januvia 100 mg po qd x 28 days for all subjects after baseline measures made
- People With Normal Glucose Tolerance: people with normal glucose tolerance
  Januvia (sitagliptin phosphate) : Januvia 100 mg po qd x 28 days for all subjects after baseline measures made
Period: Overall Study
Arm/Group | People With Impaired Fasting Glucose | People With Normal Glucose Tolerance
Started | 11 | 15
Completed | 10 | 13
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | People With Impaired Fasting Glucose | People With Normal Glucose Tolerance | Total
Number analyzed (Participants) | 11 | 15 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 15 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (2.3) | 58 (1.6) | 59 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Endogenous Glucose Production
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | People With Impaired Fasting Glucose | People With Normal Glucose Tolerance
Number analyzed (Participants) | 10 | 13
mg/kg/min
  Baseline | 1.47 (0.08) | 1.46 (0.05)
  Day 28 | 1.44 (0.04) | 1.37 (0.07)

2. Primary Outcome: Change in Insulin Secretion
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Impaired Fasting Glucose | Normal Glucose Tolerance
Number analyzed (Participants) | 10 | 13
pmol/l
  Baseline | 104 (15) | 97 (6)
  28 Days | 75 (8) | 71 (7)

3. Secondary Outcome: Insulin Secretion in Response to Oral vs. IV Glucose
Time Frame: Baseline
Population: Despite significant efforts to recover the data, data for this outcome measure could not be obtained and is not available.
Arm/Group | Impaired Fasting Glucose | Normal Glucose Tolerance
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Baseline and Change in Hormones, Substrates and Insulin Action: C-peptide
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Impaired Fasting Glucose | Normal Glucose Tolerance
Number analyzed (Participants) | 10 | 13
nmol/l
  Baseline | 0.8 (0.05) | 0.7 (0.07)
  Day 28 | 0.9 (0.03) | 0.7 (0.07)

5. Secondary Outcome: Baseline and Change in Hormones, Substrates and Insulin Action: Glucagon
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: ng/l
Arm/Group | Impaired Fasting Glucose | Normal Glucose Tolerance
Number analyzed (Participants) | 10 | 13
ng/l
  Baseline | 62 (2.8) | 63 (4.3)
  Day 28 | 61 (3.1) | 66 (4.0)

6. Secondary Outcome: Baseline and Change in Hormones, Substrates and Insulin Action: GLP-1
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Impaired Fasting Glucose | Normal Glucose Tolerance
Number analyzed (Participants) | 10 | 13
pmol/l
  Baseline | 7.5 (3.6) | 3.4 (0.7)
  Day 28 | 8.3 (2.6) | 5.4 (1.2)

7. Secondary Outcome: Baseline and Change in Hormones, Substrates and Insulin Action: Lactate
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Impaired Fasting Glucose | Normal Glucose Tolerance
Number analyzed (Participants) | 10 | 13
mmol/l
  Baseline | 0.4 (0.03) | 0.3 (0.03)
  Day 28 | 0.4 (0.09) | 0.4 (0.04)

8. Secondary Outcome: Baseline and Change in Hormones, Substrates and Insulin Action: FFA
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | Impaired Fasting Glucose | Normal Glucose Tolerance
Number analyzed (Participants) | 10 | 13
umol/l
  Baseline | 604 (30) | 610 (60)
  Day 28 | 631 (51) | 547 (44)

9. Secondary Outcome: Baseline and Change in Hormones, Substrates and Insulin Action: Glycerol
Time Frame: Baseline and 28 days
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | Impaired Fasting Glucose | Normal Glucose Tolerance
Number analyzed (Participants) | 10 | 13
umol/l
  Baseline | 91 (6) | 85 (7)
  Day 28 | 93 (6.5) | 85 (5.7)

ADVERSE EVENTS:
Arm/Group | People With Impaired Fasting Glucose | People With Normal Glucose Tolerance
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 0/11 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No